CLINICAL TRIAL: NCT03026894
Title: Association of Occlusal Force Distribution and Bone Resorption in Implant Supported Overdentures
Brief Title: Association of Force Distribution and Bone Resorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PG012-2014A
Record Dates: First submitted 2017-01-09; First posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Bone Resorption
MeSH Terms: conditions — Bone Resorption | interventions — Radiography, Panoramic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CD group (Active Comparator): Panoramic Radiographs and T-Scan III occlusal system
  Interventions: Radiation: Panoramic Radiograph; Device: T-Scan III occlusal system
- IOD group (Active Comparator): Panoramic Radiographs and T-Scan III occlusal system
  Interventions: Radiation: Panoramic Radiograph; Device: T-Scan III occlusal system

INTERVENTIONS:
Radiation: Panoramic Radiograph — Measurement of bone resorption
Device: T-Scan III occlusal system — Recording percentage of force in maximum intercuspation

SUMMARY:
To investigate the residual ridge resorption at anterior and posterior maxillary and posterior mandibular ridges among conventional complete dentures and implant overdenture wearers, and determine its association with the relative occlusal forces distribution, treatment groups and other patient variables.

DETAILED DESCRIPTION:
A total of forty-six edentulous patients participated in this clinical study divided into two groups as following; complete denture group (CD) consists of 23 patients wearing conventional complete dentures and another Implant overdenture group (IOD) consists of 23 patients wearing mandibular complete overdenture with 2 implants. Two panoramic radiographs at baseline and in a follow-up to 7 years were used to measure the ratio of bone changes between the anatomical bone area and the reference area in the maxillary and the mandibular ridges. The occlusal contacts percentage of force in maximum intercuspation anteriorly and posteriorly were recorded for both groups by using T-Scan III system.

Oral and written information in English or Malay language, regarding the study, was provided and written consent obtained before enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Patients wearing mandibular IODs opposing conventional maxillary CDs.
* Patients wearing conventional maxillary and mandibular CDs.
* Clearly visible anatomic landmarks of the panoramic radiography image.

Exclusion Criteria:

* Patients with a history of temporomandibular joint dysfunction.

Ages: 49 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-11; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Residual ridge resorption | 7 years
  To estimate residual ridge resorption in patients wearing implant overdentures and complete dentures using area index radiography method.

SECONDARY OUTCOMES:
Occlusal force distribution | 1 year
  To measure the percentage of occlusal force distribution in patients wearing implant overdentures and complete dentures using T-scan III occlusal analysis device.

IPD SHARING:
Plan to Share IPD: No